CLINICAL TRIAL: NCT02248415
Title: Administration of Warm Blood Cardioplegia With or Without Roller Pump; a Randomized Controlled Trial.
Brief Title: Administration of Warm Blood Cardioplegia With or Without Roller Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Mizja M. Faber, MSc, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL40355
Record Dates: First submitted 2014-08-25; First posted 2014-09-25 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Disease
Keywords: Cardioplegic Solutions; Myocardial Ischemia
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia | interventions — Intensive Care Units; Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No pump group (Experimental): Blood cardioplegia administration without roller pump
  Interventions: Other: No pump; Other: Blood sample collection: after induction of anaesthesia (T0); Other: Blood sample collection: after arrival at the ICU (T1); Other: Blood sample collection: 4 hours in ICU (T2); Other: Blood sample collection: the first postoperative day (T3)
- Pump group (Other): Blood cardioplegia administration with roller pump
  Interventions: Other: Pump; Other: Blood sample collection: after induction of anaesthesia (T0); Other: Blood sample collection: after arrival at the ICU (T1); Other: Blood sample collection: 4 hours in ICU (T2); Other: Blood sample collection: the first postoperative day (T3)

INTERVENTIONS:
Other: No pump — In the no pump group blood cardioplegia was delivered using the arterial line pressure, created by the arterial centrifugal pump of the cardiopulmonary bypass system. Blood cardioplegia flow depended on the difference between arterial line pressure and aortic root pressure.
  Arms: No pump group
Other: Pump — In the pump group blood cardioplegia was delivered using a roller pump. The blood cardioplegia flow was given at 200 mL/min.
  Arms: Pump group
Other: Blood sample collection: after induction of anaesthesia (T0) — The following biomarkers were analysed: TnT-hs, H-FABP, NT-pro-BNP and CRP.
Other: Blood sample collection: after arrival at the ICU (T1) — The following biomarkers were analysed: TnT-hs, H-FABP, NT-pro-BNP and CRP.
Other: Blood sample collection: 4 hours in ICU (T2) — The following biomarkers were analysed: TnT-hs, H-FABP, NT-pro-BNP and CRP.
Other: Blood sample collection: the first postoperative day (T3) — The following biomarkers were analysed: TnT-hs, H-FABP, NT-pro-BNP and CRP.

SUMMARY:
The aim of this study is to compare the effect of warm blood cardioplegia administration with and without roller pump on perioperative myocardial injury, reflected by postoperative biomarker release, in patients undergoing coronary artery bypass grafting (CABG) with a minimal extracorporeal circuit (MECC).

DETAILED DESCRIPTION:
Patients Sixty-eight patients undergoing elective coronary bypass surgery with a MECC system were consecutively enrolled and randomized into a no pump group (blood cardioplegia administration without roller pump) or pump group (blood cardioplegia administration with roller pump). Exclusion criteria were: previous cardiac surgery, scheduled surgery with less than 3 distal anastomoses, left ventricular ejection fraction <45%, chronic renal failure (defined by preoperative creatinine >177 µmol/L) and aortic insufficiency ≥ grade 1. The medical ethics committee of the St. Antonius Hospital approved this study and written informed consent was obtained for each patient prior to the surgical procedure.

Administration of blood cardioplegia In all patients warm blood cardioplegia was administered via the aortic root immediately after aortic cross-clamping. Warm blood cardioplegia consisted of oxygenated blood with added Potassium Chloride/Magnesium Sulphate (KCl/Mg SO4; Pharmacy Catharina Hospital, Eindhoven, The Netherlands: K+ 1.7 mmol/mL, Cl- 1.7 mmol/mL, Mg2+ 0.17 mmol/mL en SO4- 0.17 mmol/mL). An infusion pump was used for the addition of KCl/Mg SO4. Dosage was based on a blood cardioplegia flow of 200 mL/min and adjusted according to the following protocol: the initial dose of KCl/MgSO4 was 5.7 mmol/min (= 6.7 mL), the second dose was 3.4 mmol/min (= 4 mL) and subsequent doses were 2.6 mmol/min (= 3 mL). Each dose was given over a period of 2 minutes. Every 15 minutes the administration of blood cardioplegia was repeated. In case of recurring ECG activity, blood cardioplegia was given with aberrant intervals.

In the no pump group blood cardioplegia was delivered using the arterial line pressure, created by the arterial centrifugal pump of the cardiopulmonary bypass system. Blood cardioplegia flow depended on the difference between arterial line pressure and aortic root pressure. In the pump group blood cardioplegia was delivered using a roller pump. The blood cardioplegia flow was given at 200 mL/min.

Blood sample collection and analyses Blood was collected in EDTA tubes (6 mL) at baseline after induction of anaesthesia (T0), after arrival at the ICU (T1), 4 hours in ICU (T2) and at the first postoperative day (T3). Blood samples were fractionated by centrifuging 1500-2000 x g for 15 min. Plasma was collected and stored at -80°C until analysis. The following biomarkers were analysed: Troponin T high sensitive (TnT-hs), Heart-type Fatty Acid Binding Protein (H-FABP), N-terminal brain natriuretic peptide (NT-pro-BNP) and C-reactive protein (CRP).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective coronary artery bypass grafting
* Scheduled surgery with less than 3 distal anastomoses

Exclusion Criteria:

* Previous cardiac surgery
* Left ventricular ejection fraction <45%
* Chronic renal failure (defined by preoperative creatinine >177 µmol/L)
* Aortic insufficiency ≥ grade 1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Troponin T high sensitive (TnT-hs) (ng/L) | Change from baseline to the first postoperative day
Heart-type Fatty Acid Binding Protein (hFABP) (ng/mL) | Change from baseline to the first postoperative day
N-terminal brain natriuretic peptide (NT-pro-BNP) (ng/mL) | Change from baseline to the first postoperative day
C-reactive protein (CRP) (μg/mL) | Change from baseline to the first postoperative day

SECONDARY OUTCOMES:
Blood cardioplegia flow during blood cardioplegia delivery (mL/min) | Intraoperative
Arterial line pressure during blood cardioplegia delivery (mmHg) | Intraoperative
Blood cardioplegia line pressure during blood cardioplegia delivery (mmHg) | Intraoperative
Aortic root pressure during blood cardioplegia delivery (mmHg) | Intraoperative
Post-operative myocardial infarction | 30-days
Inotropic support (hours) | 30-days
TIA/CVA | 30-days
Pneumonia | 30-days
Renal failure | 30-days
  Creatine>177 μmol/l/l
Re-thoracotomy | 30-days
Atrial fibrillation | 30-days
Length of ICU stay (hours) | 30-days
Length of hospital stay (days) | 30-days

CONTACTS AND LOCATIONS:
Overall Officials: Mizja Faber, Faber, Principal Investigator — mizjafaber@heartbeat5.nl
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands